CLINICAL TRIAL: NCT01658943
Title: Randomized Phase II Clinical Trial of AZD6244 Hydrogen Sulfate (NSC-748727) and MK-2206 (NSC-749607) vs mFOLFOX in Patients With Metastatic Pancreatic Cancer After Prior Chemotherapy
Brief Title: Selumetinib and Akt Inhibitor MK2206 or mFOLFOX Therapy Comprising Oxaliplatin and Fluorouracil in Treating Patients With Metastatic Pancreatic Cancer Previously Treated With Chemotherapy
Acronym: S1115
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01993; NCI-2012-01993 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S1115; CDR0000737878; S1115 (Other: SWOG); S1115 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2015-07

CONDITIONS: Pancreatic Acinar Cell Carcinoma; Pancreatic Ductal Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — MK 2206; Fluorouracil; dehydroftorafur; Oxaliplatin; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (mFOLFOX regimen) (Experimental): Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and fluorouracil IV over 46-48 hours on days 1-2 and 15-16.
  Interventions: Drug: Fluorouracil; Drug: Oxaliplatin
- Arm II (Akt inhibitor MK2206 and selumetinib) (Experimental): Patients receive Akt inhibitor MK2206 PO on days 1, 8, 15, and 22, and selumetinib PO daily on days 1-28.
  Interventions: Drug: Akt Inhibitor MK2206; Drug: Selumetinib

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
  Arms: Arm II (Akt inhibitor MK2206 and selumetinib)
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Actino-Hermal; Adrucil; Arumel; Cytosafe; Efudex; Efurix; Fiverocil; Fluoro Uracil; Fluoroplex; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Flurox; Ribofluor; Ro 2-9757; Ro-2-9757; Timazin
  Arms: Arm I (mFOLFOX regimen)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
  Arms: Arm I (mFOLFOX regimen)
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244
  Arms: Arm II (Akt inhibitor MK2206 and selumetinib)

SUMMARY:
This randomized phase II trial studies how well selumetinib and Akt inhibitor MK2206 work compared to modified fluorouracil, leucovorin calcium, and oxaliplatin (mFOLFOX) therapy in treating patients with metastatic pancreatic cancer previously treated with chemotherapy. Selumetinib and Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as oxaliplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet know whether selumetinib and Akt inhibitor MK2206 are more effective than oxaliplatin and fluorouracil in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess overall survival in patients with metastatic pancreatic cancer treated with the combination of AZD6244 hydrogen sulfate (selumetinib) and MK-2206 (Akt inhibitor MK2206) compared to those treated with mFOLFOX.

SECONDARY OBJECTIVES:

I. To assess the frequency and severity of toxicity associated with the combination of AZD6244 hydrogen sulfate and MK-2206 compared to those with mFOLFOX in this patient population.

TERTIARY OBJECTIVES:

I. To assess progression free survival (PFS) in patients with metastatic pancreatic cancer treated with the combination of AZD6244 hydrogen sulfate and MK-2206 compared to those treated with mFOLFOX.

II. To assess objective tumor response in the subset of patients with measurable disease (confirmed and unconfirmed complete and partial response) in patients with metastatic pancreatic cancer treated with the combination of AZD6244 hydrogen sulfate and MK-2206 compared to those treated with mFOLFOX.

III. To bank tissue and blood for future translational medicine studies.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oxaliplatin intravenously (IV) over 2 hours on days 1 and 15 and fluorouracil IV over 46-48 hours on days 1-2 and 15-16 (mFOLFOX).

ARM II: Patients receive Akt inhibitor MK2206 orally (PO) on days 1, 8, 15, and 22, and selumetinib PO daily on days 1-28.

In all arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma; patients with endocrine or neuroendocrine tumors, lymphoma of the pancreas, or ampullary cancer are not eligible
* Patients must have distant metastatic disease; patients with macroscopic residual disease post-resection as the only site of disease are not eligible; patient must not have clinically significant ascites (defined as requiring paracentesis) or have brain metastases
* Patients must have received one line, and no more than one line, of prior gemcitabine-based chemotherapy for advanced/metastatic pancreatic cancer and must have documentation of metastatic disease progression while on this treatment; documented disease progression must occur within 42 days of the last treatment; OR

  * For patients who received one line of gemcitabine-based chemotherapy for treatment in the adjuvant setting, recurrence to a metastatic site must be documented by imaging studies within 6 months of completing chemotherapy; chemoradiation as part of adjuvant treatment is acceptable; if the patient received one line of adjuvant gemcitabine-based treatment and had disease recurrence after 6 months of completing chemotherapy, patients will only be eligible after failing one additional line of gemcitabine-based chemotherapy used to treat the metastatic disease
* Patients must have measurable and/or non-measurable disease; x-rays, scans. or physical examinations for assessment of measurable disease must have been completed within 28 days prior to registration; x-rays, scans, or other tests for assessment of non-measurable disease must have been completed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients must have completed systemic therapy at least 14 days prior to registration, any surgical procedure must have been performed at least 14 days prior to registration, and radiation therapy must be completed at least 7 days prior to registration; patients must have recovered to =< grade 1 from any of the effects of prior therapies or procedures
* Patients must not plan to receive concurrent chemotherapy, radiotherapy, agents known to prolong corrected QT (QTc) interval, or agents known to be strong inducers or inhibitors of cytochrome P450 3A4/5 (CYP3A4/5) or cytochrome P450 1A2 (CYP1A2)
* Patient must not have received prior treatment with fluorouracil, irinotecan, leucovorin calcium, and oxaliplatin (FOLFIRINOX), FOLFOX, oxaliplatin-based chemotherapy, mitogen-activated protein kinase (MEK) inhibitors, phosphoinositide-3-kinase (PI3K) inhibitors, or protein kinase B (AKT) inhibitors
* Zubrod performance status of 0-1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9.0 g/dL
* Patients must have adequate kidney function as evidenced by at least ONE of the following:

  * Serum creatinine =< 1.5 mg/dL within 14 days prior to registration
  * Calculated creatinine clearance >= 60 mL/min; the serum creatinine value used in the calculation must have been obtained within 14 days prior to registration
* Total bilirubin =< 1.5 times institutional upper limit of normal(IULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 2.5 times IULN
* Patients must have an albumin level >= 3.0 g/dL within 14 days prior to registration
* Patients must have an International Normalized Ratio (INR) =< 1.5 times IULN within 14 days prior to registration
* Patients must have an electrocardiogram (ECG) within 14 days prior to registration; patients must have QTcF (by Fridericia's calculation) =< 450 msec (male) or =< 470 msec (female)
* Patients with baseline neuropathy must be =< grade 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v 4.0
* Patients must not have uncontrolled diarrhea or active infection requiring antibiotics and be fully recovered from any previous serious infections within 7 days prior to registration
* Patients must be able to swallow tablets and capsules
* Patients with diabetes must be well controlled with fasting glucose =< grade 1 according to CTCAE v 4.0 within 14 days prior to registration
* Patients with history of congestive heart failure must have an ejection fraction >= 55% within 14 days prior to registration
* Patients must not have any of the following: uncontrolled hypertension, acute coronary syndrome within 6 months prior to registration, poorly controlled angina, New York Heart Association class II-IV heart failure, prior or current cardiomyopathy, atrial fibrillation, or severe valvular heart disease
* Patients must not have a current or past history of central serous retinopathy, retinal vein occlusion, retinal detachment, or have uncontrolled glaucoma (irrespective of intraocular pressure [IOP])
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for five years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method during the study plus at least 16 weeks after last dose; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Prestudy history and physical must be obtained within 28 days prior to registration
* Sites must seek additional patient consent for the future use of specimens
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — SWOG Cancer Research Network
Locations (534):
- United States (534):
  - The University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - East Bay Medical Oncology Hematology Medical Associates Inc-Pleasant Hill, Pleasant Hill, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Baptist Cancer Institute, Jacksonville, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Central Illinois CCOP, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan St. Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Cancer Center of Acadiana, Lafayette, Louisiana
  - DeSoto Regional Health System, Mansfield, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Cancer Control Consortium CCOP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Akron General Medical Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Oncology Inc, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Cancer Research Foundation, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Danville Hematology Oncology, Danville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative of Puget Sound Oncology Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Chung V, McDonough S, Philip PA, Cardin D, Wang-Gillam A, Hui L, Tejani MA, Seery TE, Dy IA, Al Baghdadi T, Hendifar AE, Doyle LA, Lowy AM, Guthrie KA, Blanke CD, Hochster HS. Effect of Selumetinib and MK-2206 vs Oxaliplatin and Fluorouracil in Patients With Metastatic Pancreatic Cancer After Prior Therapy: SWOG S1115 Study Randomized Clinical Trial. JAMA Oncol. 2017 Apr 1;3(4):516-522. doi: 10.1001/jamaoncol.2016.5383. PMID 27978579

RESULTS

PARTICIPANT FLOW:
Groups:
- mFOLFOX: Patients receive 85 mg/m^2 oxaliplatin IV over 2 hours on days 1 and 15 and 2,400 mg/m^2 fluorouracil IV over 46-48 hours on days 1-2 and 15-16. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
- MK2206 and Selumetinib: Patients receive 135 mg MK2206 PO on days 1, 8, 15, and 22, and 100 mg selumetinib PO daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | mFOLFOX | MK2206 and Selumetinib
Started | 70 | 67
Eligible | 63 | 58
Eligible and Began Protocol Therapy | 62 | 58
Completed | 0 | 0
Not Completed | 70 | 67
Not completed — Adverse Event | 6 | 13
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Progression/Relapse | 39 | 40
Not completed — Death | 4 | 2
Not completed — not protocol specified | 4 | 1
Not completed — Not eligible | 7 | 9
Not completed — Withdrew prior to beginning protocol Tx | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and analyzable patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFOX | MK2206 and Selumetinib | Total
Number analyzed (Participants) | 62 | 58 | 120
Age, Continuous [Median (Full Range); unit: years] | 65.6 [34.2 to 82.8] | 69.4 [54.2 to 88.0] | 67.3 [34.2 to 88.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 23 | 63
  Male | 22 | 35 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 59 | 57 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 7 | 4 | 11
  White | 50 | 49 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Prior Systemic Therapy [Number; unit: participants]
  4 months or less | 23 | 22 | 45
  more than 4 months | 39 | 36 | 75
Liver Metastasis [Number; unit: participants]
  Yes | 39 | 43 | 82
  No | 23 | 15 | 38

OUTCOME MEASURES:

1. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary.
Measure: Number; unit: Participants
Arm/Group | mFOLFOX | MK2206 and Selumetinib
Number analyzed (Participants) | 62 | 57
Participants
  Abdominal pain | 1 | 0
  Alanine aminotransferase increased | 0 | 4
  Alkaline phosphatase increased | 0 | 2
  Anemia | 2 | 3
  Anorexia | 1 | 1
  Aspartate aminotransferase increased | 0 | 3
  Blood bilirubin increased | 1 | 0
  Cognitive disturbance | 0 | 1
  Dehydration | 1 | 6
  Device related infection | 1 | 0
  Diarrhea | 4 | 4
  Edema face | 0 | 1
  Encephalopathy | 0 | 1
  Erythema multiforme | 0 | 1
  Erythroderma | 0 | 1
  Fatigue | 8 | 7
  Generalized muscle weakness | 0 | 1
  Hepatic failure | 0 | 1
  Hyperglycemia | 1 | 7
  Hypertension | 2 | 5
  Hypokalemia | 1 | 1
  Hypomagnesemia | 1 | 0
  Hyponatremia | 1 | 4
  Hypophosphatemia | 0 | 1
  Hypotension | 1 | 1
  Hypoxia | 0 | 1
  Left ventricular systolic dysfunction | 0 | 1
  Lung infection | 1 | 1
  Lymphocyte count decreased | 8 | 0
  Mucositis oral | 1 | 4
  Multi-organ failure | 0 | 1
  Nausea | 3 | 0
  Neoplasms benign, malignant and unspecified | 0 | 2
  Neutrophil count decreased | 4 | 0
  Platelet count decreased | 1 | 0
  Rash acneiform | 0 | 5
  Rash maculo-papular | 0 | 7
  Skin infection | 0 | 1
  Soft tissue infection | 0 | 1
  Stevens-Johnson syndrome | 0 | 1
  Syncope | 0 | 1
  Vomiting | 3 | 1
  Weight loss | 1 | 0
  White blood cell decreased | 2 | 0

2. Primary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 3 years
Population: Eligible and analyzable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | mFOLFOX | MK2206 and Selumetinib
Number analyzed (Participants) | 62 | 58
months | 6.7 [6.0 to 8.3] | 3.9 [3.5 to 4.6]
Statistical Analysis 1: Comparison: mFOLFOX vs MK2206 and Selumetinib; Test type: Superiority or Other; p = 0.15, Log Rank

3. Other Pre Specified Outcome: Progression-free Survival
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression free are censored at date of last contact.
Time Frame: Up to 3 years
Population: Eligible and analyzable patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | mFOLFOX | MK2206 and Selumetinib
Number analyzed (Participants) | 62 | 58
months | 2.0 [1.8 to 2.9] | 1.9 [1.8 to 2.1]

4. Other Pre Specified Outcome: Objective Response Rate
Description: Confirmed response (CR) is two or more objective statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Partial response (PR) is two or more objective statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration. Unconfirmed CR is one objective status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one objective status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 3 years
Population: All eligible and analyzable patients with measurable disease.
Measure: Number; unit: participants
Arm/Group | mFOLFOX | MK2206 and Selumetinib
Number analyzed (Participants) | 57 | 55
participants
  Partial Response | 4 | 0
  Unconfirmed Partial Response | 1 | 1
  Stable/No response | 14 | 12
  Increasing disease | 29 | 34
  Symptomatic Deterioration | 3 | 2
  Assessment Inadequate | 6 | 6

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Eligible patients who received any treatment and were assessed for adverse events are included in the adverse event summaries.
Arm/Group | mFOLFOX | MK2206 and Selumetinib
Serious Adverse Events (participants affected / at risk) | 2/62 | 37/57
Other Adverse Events (participants affected / at risk) | 56/62 | 53/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX (N=62) | MK2206 and Selumetinib (N=57)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 3
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Fever (General disorders) | 0 | 2
General disorders and admin site conditions - Other (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Investigations-Other (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 10
Cognitive disturbance (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 4
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 3
Visceral arterial ischemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX (N=62) | MK2206 and Selumetinib (N=57)
Anemia (Blood and lymphatic system disorders) | 26 | 17
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 26 | 14
Ascites (Gastrointestinal disorders) | 1 | 3
Bloating (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 25 | 8
Diarrhea (Gastrointestinal disorders) | 23 | 17
Dry mouth (Gastrointestinal disorders) | 0 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Flatulence (Gastrointestinal disorders) | 1 | 4
Mucositis oral (Gastrointestinal disorders) | 8 | 12
Nausea (Gastrointestinal disorders) | 39 | 25
Vomiting (Gastrointestinal disorders) | 21 | 21
Chills (General disorders) | 2 | 10
Edema face (General disorders) | 0 | 6
Edema limbs (General disorders) | 6 | 9
Fatigue (General disorders) | 39 | 25
Fever (General disorders) | 4 | 6
Pain (General disorders) | 4 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 6
Alanine aminotransferase increased (Investigations) | 9 | 17
Alkaline phosphatase increased (Investigations) | 18 | 13
Aspartate aminotransferase increased (Investigations) | 13 | 20
Blood bilirubin increased (Investigations) | 5 | 3
Creatinine increased (Investigations) | 3 | 9
Investigations-Other (Investigations) | 4 | 4
Lymphocyte count decreased (Investigations) | 15 | 8
Neutrophil count decreased (Investigations) | 12 | 1
Platelet count decreased (Investigations) | 21 | 6
Weight loss (Investigations) | 13 | 6
White blood cell decreased (Investigations) | 13 | 1
Anorexia (Metabolism and nutrition disorders) | 25 | 20
Dehydration (Metabolism and nutrition disorders) | 7 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 20 | 22
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 | 17
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 7
Hypokalemia (Metabolism and nutrition disorders) | 11 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatremia (Metabolism and nutrition disorders) | 10 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 6
Dizziness (Nervous system disorders) | 4 | 10
Dysgeusia (Nervous system disorders) | 8 | 8
Headache (Nervous system disorders) | 6 | 2
Paresthesia (Nervous system disorders) | 7 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 29 | 4
Anxiety (Psychiatric disorders) | 5 | 4
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 8
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 18
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 3
Hypertension (Vascular disorders) | 8 | 7
Hypotension (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less